CLINICAL TRIAL: NCT05959928
Title: Temperature Telemonitoring for Hospital at Home (HaH) Patients
Brief Title: Continuous Temperature Telemonitoring of Patients With COVID-19 and Other Infectious Diseases in Hospital at Home Using Viture
Acronym: Viture
Status: Completed | Type: Observational
Sponsor: Vitio Medical S.L. (Industry)
Collaborators: Hospital of Navarra (Other); NavarraBiomed Biomedical Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: 859/20/EC
Record Dates: First submitted 2023-07-20; First posted 2023-07-25 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: COVID-19; Infectious Disease; Tract Infection, Urinary; Bacteremia; Respiratory Infection; Cellulitis
Keywords: Continuous body temperature monitoring; Hospital at Home; Telemonitoring; Remote Patient Monitoring; Virtual wards; Fever detection; Infectious diseases; Telemedicine; Telehealth; COVID-19; Real-time data
MeSH Terms: conditions — COVID-19; Communicable Diseases; Urinary Tract Infections; Bacteremia; Respiratory Tract Infections; Cellulitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hospital at Home patients
  Interventions: Device: Continuous wearable thermometer placed on patient's armpit to monitor body temperature remotely

INTERVENTIONS:
Device: Continuous wearable thermometer placed on patient's armpit to monitor body temperature remotely — The HaH team will place Viture Device on the patient's armpit and train the patient and/or caregiver. They will ask to complete control STMs between 3 and 6 times a day on the same arm where the Viture Device is placed and record the measuring data in the Home data collection notebook (HDCN)

SUMMARY:
The aim of this cohort study is to validate Viture®, a continuous temperature telemonitoring system, evaluating the level of agreement with a standard commercially available digital axillary thermometer. The study also aims to evaluate the safety and comfort of the system and to evaluate the impact that the introduction of Viture has on the health care practice of a HaH unit. Furthermore, the advantages of Viture compared to the standard method will be evaluated.

DETAILED DESCRIPTION:
Body temperature is a key vital sign in the follow-up of patients admitted to Hospital at Home (HaH) units with COVID-19 and other infectious diseases. Continuous telemonitoring of temperature can lead to earlier detection of fever and patient deterioration that facilitates early decision making.

In the first day of the study, the patients will be given a study kit of Viture System with the following content:

* Viture Device.
* Digital reference thermometer for control Spot Temperature Measurements (STMs)
* Smartphone with Viture Mobile App installed.
* Device user manual in quick guide format.
* Home data collection notebook (HDCN)

The HaH team will place Viture Device on the patient and train the patient and/or caregiver. They will ask patients to complete control STMs between 3 and 6 times a day on the same arm where the Viture Device is placed and record the measuring data in the HDCN.

In the case that the bracelet is removed, or the patient experience discomfort, they will be asked to fill in the incident in the HDCN. Mild incidents are considered skin alterations such as redness and chafing and severe incidents are considered hematomas and ulcers.

The HaH team on duty will collect all Viture notifications, registering the date, time, and follow-up for each febrile episode. The patient and/or caregiver could be contacted to request a control STM.

A statistical analysis of agreement between the digital reference thermometer (Gold standard) and Viture will be carried out. The non-parametric Wilcoxon signed rank test will be used to evaluate the average agreement between the two methods, and the Bland Altman method will be used to evaluate the agreement between individual measurements. Both analyses will be validated with a 95% confidence interval.

To explore the true potential of Viture, an analysis of the febrile episodes experienced by patients during the clinical study will be performed. Febrile episodes will be characterized by their maximum temperature and duration. To assess the impact of Viture notifications, the data registered on the follow-up of febrile episodes will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* be more than 18 years old.
* to be able to legally give informed consent.
* not to have limitations to the use of the Viture Device due to their physical conditions or interference with other devices.

Exclusion Criteria:

* To be monitored for less than 2 days.
* To have less than 4 valid control Spot Temperature Measurements (STM). A valid control STM is considered a temperature measured with the reference thermometer that has a simultaneous (within 1 minute) Viture Temperature Measurement (VTM)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years old who have been admitted to Hospital at Home (HaH) units with COVID-19 and other infectious diseases.
Sampling Method: Probability Sample
Enrollment: 208 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2021-06-02 (Actual); Study Completion 2021-06-02 (Actual)

PRIMARY OUTCOMES:
Verify that, under normal conditions of use, the performance of Viture for body temperature measurement is equivalent to the devices used in the standard practice. | 3 measurements per day
  Comparison between the temperatures recorded remotely by Viture and a control digital thermometer used in the follow-up of patients in Hospital at Home, both COVID-19 patients and patients with other diseases who benefit from body temperature monitoring.

SECONDARY OUTCOMES:
Evaluate the safety, usability and comfort of Viture Device | Through study completion, an average of 5 days
  Record usability experience and negative sensations expressed by users due to the use of Viture, such as discomfort or skin irritation in the area where the device is placed.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Ruiz Castellano, MD, Principal Investigator — Hospital of Navarra
Locations (1):
- Hospital Universitario de Navarra, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No